CLINICAL TRIAL: NCT00444301
Title: Investigating Pain in Heart Failure Patients
Brief Title: Pain Assessment, Incidence & Nature in Heart Failure
Acronym: PAIN-HF
Status: Completed | Type: Observational
Sponsor: PC-HEART (Other)
Collaborators: Mayday Fund (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sarah Goodlin MD/ Principal Investigator, Patient-centered Education and Research
Other Study IDs: 06-117PCER
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Heart Diseases
Keywords: Heart failure; Pain; Symptoms; Advanced heart failure; Pain frequency, severity, location, treatments; Shortness of breath, anxiety, depression, cognitive function; Social support, other conditions and illnesses
MeSH Terms: conditions — Heart Diseases; Heart Failure; Pain; Dyspnea; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart failure, a chronic illness afflicting 5 million persons in the United States is known to cause shortness of breath and fatigue, yet at least half of persons with heart failure also report the presence of pain.

The cause of pain for these persons is not clear. PAIN-HF (Pain Assessment, Incidence & Nature in Heart Failure), conducted through the Palliative Care-Heart Failure Education And Research Trials (PC-HEART) collaborative will identify the prevalence of pain, its location, severity and impact on activities and the possible causes of pain in persons living with heart failure. The study will also try to understand relationships between other problems and pain, as well as what treatments are given to reduce pain.

Understanding sources of pain and its characteristics is the first step in helping health care providers better manage pain and related problems in persons with heart failure.

DETAILED DESCRIPTION:
Subjects will be recruited via physicians and nurses providing their care in clinical sites who are members of PC-HEART. PC-HEART is a volunteer collaborative with clinician-investigators at 60 sites nationally that include hospice organizations and heart failure providers in academic, Health Maintenance Organization (HMO) and community settings. Our goal will be to enroll 400 patients with 135 in hospice care and 265 in outpatient settings (a mix of HMO, community practice, VA, and academic centers) who are members of the Palliative Care- Heart Failure Education And Research Trials (PC-HEART) collaborative. We will strive for broad representation of patients living in the community with about one-third African American patients (who often present for initial treatment with advanced heart failure) and at least one-half elderly (who have high prevalence of both pain and heart failure).

We will use standardized tools to survey patients, as follows:

Pain & other symptoms (Assessed at enrollment and one-two weeks later):

Memorial Symptom Assessment Scale- HF (MSAS-HF) Short-form McGill pain questionnaire (SF-MPQ) Brief Pain Inventory (BPI)

Heart-failure specific measures (Assessed at Enrollment):

Kansas City Cardiomyopathy Questionnaire (KCCQ)

Psycho-social situation & cognitive function (Assessed at Enrollment):

Physicians Health Questionnaire depression screen (PHQ-9) Mini-cog Social functioning: ENRICHD Social Support Inventory (ESSI) , The Short Physical Performance Battery (SPPB) will be collected on 1/2 of subjects Clinical Data (from medical record) Patient's medical condition: Charleson Comorbidity Scale, prior diagnosis of Diabetes Mellitus, Cancer, Chronic lung disease, Coronary Artery Disease, Cirrhosis.

Known painful conditions (osteoarthritis, chronic back pain, CAD with angina, neuropathy, others) Physical examination: Jugular Venous Pressure (as per NIH trial standards: base of neck, ½ way up, jaw level), edema (+1 (0-1/4" depression), +2 (1/4-1/2"), +3 (1/2-1"), +4 (>1")), Blood pressure, Respiratory rate, Heart rate & rhythm Echocardiogram data: Date of most recent Echocardiogram, LVEF, LVDD, LA dimension, presence of valvular disease & measure of severity (for example, if aortic stenosis then valve area, if mitral regurgitation then 1+-4+) Laboratory data: BUN, CR, Na+, HgB, BNP, hemoglobin

Demographic Data Age, Sex, Race & ethnic identification, Marital Status, Living situation (alone, with family, with other person), employment status (employed, self-employed, retired, unemployed due to disability), highest level of education, religious affiliation, annual household income, insurance (none, Medicare, Medicaid, Veterans Administration, Kaiser, other Health Maintenance Organization, private fee for service).

Medications & Treatment (Assessed at Enrollment and 1-2 weeks later) Heart Failure medications: ACEI, ARB, β-blocker, digoxin, spironolactone, eplerenone, loop diuretics, nesiritide, inotropes, warfarin Analgesics: NSAIDs, Cox-2 inhibitors, Aspirin, Acetaminophen, Tramadol, Opioids Antidepressants: SSRI, Tricyclics, Psychostimulants, other Topical agents: acetylsalicylate acid creams, capsaicin Physical therapy, cold, heat, other modalities Statistical Evaluation We will report frequencies of pain in total, frequencies of levels of severity & interference in activities of pain, by occasional versus frequent or constant pain, and by location with descriptive statistics. To the extent the etiology of pain is identified this will be reported with descriptive statistics. Pearson product-moment correlation coefficients, t-test and frequency statistics (Chi-square and Fisher's Exact test) will be used to evaluate associations between pain presence, severity and type and demographic and clinical variables. If possible, comparison will be made between patients without pain and those with pain using chi-square tests and t-test.

A multivariate analysis of variance will be used to assess relationship between pain and measures of heart failure severity, social support, depression and symptom distress other than pain.

Differences in Pain measures will be assessed between enrollment and the second assessment 1-2 weeks later, and changes will be correlated with changes in treatment for pain. Geographic locations of pain will be mapped using the body diagram on the BPI to identify areas of greatest frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced HF (Stage D or advanced Stage C HF) with:

   symptoms of dyspnea at rest or with minimal exertion systolic dysfunction or preserved systolic function ("diastolic heart failure") Outpatient care setting (office, clinic or home hospice).
2. Patient already receiving optimal medical therapy per ACC/AHA guidelines (ACEI or ARB + β-blocker +aldosterone antagonist) for at least 1 month or explanation of intolerance of specific medication. We will exclude those not on optimized medications with no notation of intolerance; however, we will keep a tally to quantify patients who are considered "advanced Heart Failure" but are not on recommended medications.
3. Can be awaiting LVAD, transplantation or other procedure
4. Age > 18 years and able to sign informed consent to participate

Exclusion Criteria:

1. Cognitive or other impairment which prevents accurate assessment of symptoms or ability to provide informed consent.
2. Heart failure due to recent onset of acute viral myocarditis, peripartum myocarditis.
3. Patient on hemodialysis or receiving mechanical ventilation
4. Patients receiving investigational agents or devices.
5. Patients who have received heart transplant or a destination Left Ventricular Assist Device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced heart failure
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Goodlin, MD, Principal Investigator — Patient-centered Education and Research
Locations (14):
- United States (14):
  - San Diego Hospice & Palliative Care, San Diego, California
  - Washington DC VAMC Heart Failure Clinic, Washington D.C., District of Columbia
  - Hospice of Palm Beach County, Palm Beach, Florida
  - Lifepath Hospice & Palliative care, Tampa, Florida
  - Bluhm Cardiovascular Institute, Chicago, Illinois
  - Unniversity of Kentucky, Lexington, Kentucky
  - Kaiser Mid-Atlantic States, Silver Spring, Maryland
  - Singing River Hospital System, Pascagoula, Mississippi
  - Strong Memorial Congestive Heart Failure Program, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospice of Lancaster County/The Heart Group, Lancaster, Pennsylvania
  - Caris Health Care, Knoxville, Tennessee
  - The Heart Center, Holladay, Utah
  - Capital Hospice, Falls Church, Virginia

REFERENCES:
- See also: This is the PC-HEART website — http://www.pc-heart.org